CLINICAL TRIAL: NCT05649514
Title: Objective Sleep Impairment in APOEε4/ε4 Subjects at Risk of Developing Alzheimer's Disease: Risk Factor for Cognitive Decline?
Brief Title: Sleep Impairment in Subjects at Risk of Developing Alzheimer's Disease
Acronym: WAVE-APOE4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0392
Record Dates: First submitted 2022-11-09; First posted 2022-12-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Neuropathology; Cognitive Decline; Sleep Disorder
Keywords: cognitive composite score; sleep; biomarkers; cognitive decline
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Wake Disorders | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Prodromal Alzheimer's patients
  Interventions: Procedure: Polysomnography; Behavioral: Neuropsychological assessment; Behavioral: Questionnaires on sleep and behavioural problems; Procedure: Actimetrics; Other: Biomarker assay

INTERVENTIONS:
Procedure: Polysomnography — Polysomnography will be performed for 24 hours at inclusion and 24 months
Behavioral: Neuropsychological assessment — A full neuropsychological assessment will be performed at inclusion, 12 and 24 months
Behavioral: Questionnaires on sleep and behavioural problems — Questionnaires on sleep and behavioural problems
Procedure: Actimetrics — Measurement of actimetrics for 14 days at inclusion and at 24 months
Other: Biomarker assay — Determination of the biomarkers Aβ42, Aβ40, Tau and P-Tau in blood and in the cerebrospinal fluid

SUMMARY:
Alzheimer's disease (AD) is characterised by a progressive loss of memory and cognitive function. In the early stages of AD, there is a progressive accumulation of molecules: β-amyloid peptides (Aβ) in the brain. There is a link between the accumulation of Aβ peptides and the deterioration of sleep, but current knowledge does not confirmed this link. The objective of this study is to define whether there is a link between cognitive decline and sleep disorders. If a correlation is found, this could allow earlier treatment of sleep disorders in the longer term in order to slow the development of AD.

Treatment protocols in the field of Alzheimer's disease (AD) are directed towards participants at risk of developing the disease, such as those who carry at least one ε4 allele on apolipoprotein E (APOE ε4). An individual with 2 ε4 copies has a 30-55% risk of developing AD with an age of onset around 68 years and a dose effect of the allele on risk and age of onset of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild Alzheimer's disease with a MMS between 21-30
* Without anticholinesterase and/or memantine treatment or on stable doses for at least 3 months
* No antidepressant or anxiolytic treatment or stopped for at least 15 days
* The presence of a family carer to complete neuropsychological scales, questionnaires and sleep diaries
* Signed informed consent
* Able to carry out all visits and follow study procedures
* Affiliation to the French social security system

Exclusion Criteria:

* Genetic form of alzheimer's disease
* Insufficient clinical and paraclinical information for the diagnosis of AD
* Patient living in a nursing home
* Illiteracy or inability to perform psycho-behavioural tests
* Major physical or neurosensory problems that may interfere with the tests
* Patient deprived of liberty, by judicial or administrative decision;
* Major depression according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Major protected by law;
* Short-term life-threatening conditions

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Alzheimer's Disease Cooperative Study - Preclinical Alzheimer Cognitive (ADCS-PACC) scale score | From inclusion to 24 months
  The ADCS-PACC scale will be based on scores from the Mini Mental State Examination (MMSE), the Free Recall/Indicated Recall Test, the Digit Substitution Symbol Test, the Wechsler Intelligence Scale for Adults (WAIS-IV), and the 2-minute Verbal Fluency Test

SECONDARY OUTCOMES:
Change in the Alzheimer's Disease Cooperative Study - Preclinical Alzheimer Cognitive (ADCS-PACC) scale score | From inclusion to 12 months
  The ADCS-PACC scale will be based on scores from the Mini Mental State Examination (MMSE), the Free Recall/Indicated Recall Test, the Digit Substitution Symbol Test, the Wechsler Intelligence Scale for Adults (WAIS-IV), and the 2-minute Verbal Fluency Test
Cognitive decline in ADCS-PACC composite score | At inclusion and at 12 months
  The ADCS-PACC composite score is used to assess cognitive decline
Concentration of proteins involved in Alzheimer disease | At inclusion and at 24 months
  Determination of Aβ42, Aβ40, Tau and P-Tau proteins in serum and cerebrospinal fluid
Sleep time at stage 1-2 during polysomnography | At inclusion and at 24 months
  Time spent in stage 1-2 sleep measured in hours and minutes during polysomnography
Sleep time at stage 3 during polysomnography | At inclusion and at 24 months
  Time spent in stage 3 sleep measured in hours and minutes during polysomnography
Time spent in Rapide Eye Movement (REM) sleep during polysomnography | At inclusion and at 24 months
  Time spent in REM in hours and minutes during polysomnography
Apnea Hypopnea index | At inclusion and at 24 months
  The Apnea-Hypopnea Index is calculated from the number of apneas and hypopneas per hour of sleep (AHI = number of apneas + number of hyopneas / number of hours of sleep) during polysomnography
Noctural oxygene saturation (SaO2) | At inclusion and at 24 months
  The noctural SaO2 is an average of SaO2 values taken during the night. The value is expressed as a percentage and is measured during polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Karim BENNYS, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No